CLINICAL TRIAL: NCT01329575
Title: Predicting Malignancy Using Endoluminal Ultrasound Characteristics in Mediastinal Lymph Nodes
Acronym: CT0024
Status: Completed | Type: Observational
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Centre de Recherche du Centre Hospitalier de l'Université de Montréal (Other)
Responsible Party: Sponsor
Other Study IDs: CE 11.005
Record Dates: First submitted 2011-04-04; First posted 2011-04-06 (Estimated); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Neoplasm of Mediastinal Lymph Nodes
Keywords: endoluminal ultrasound; Mediastinal LN invasion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
There is no single method to investigate mediastinal LN invasion. Hence, a patient may have to undergo several tests and procedures. Noninvasive and invasive approaches are employed. Within the invasive techniques, endoscopic ultrasonography with needle aspiration (EUS-FNA) and endobronchial ultrasonography with transbronchial needle aspiration (EBUS-TBNA) are gaining importance in mediastinal staging.5 They provide ultrasonographic images and permit needle aspiration under direct vision for cytology specimen analysis. As more evidence is being accumulated on these staging approaches, the number of cervical mediastinoscopies, considered as the gold-standard for mediastinal staging, is diminishing.

Color Doppler LN characteristics with endoluminal ultrasound (US) is only mentioned in a small number of studies and needs to be further investigated.13,14 With the good results obtained with superficial US, it seems reasonable to believe that color Doppler characteristics would increase accuracy in detecting malignancy of mediastinal LNs with endoluminal US.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer-related death in the United States with a 5-year survival rate of 15,7%.1 In lung cancer and other malignancies, such as esophageal cancer, accurate staging is essential to establish prognosis and for patient management. Staging will help determine if surgery, chemotherapy, radiation therapy, a combination of these, or a palliative approach is the most adequate.2,3

Assessment of lymph nodes (LNs) for invasion by metastasis is undertaken if patient management is influenced by a positive or negative result. In non-small cell lung cancer (NSCLC), mediastinal LN invasion by malignant cells is a critical factor to determine if a patient is considered as a surgical candidate or not.2 In esophageal cancer, LN metastasis may be found in the mediastinum, the neck and the abdomen.4 Invasion of these LNs must be considered in the selection of treatment of esophageal cancer.3,4

There is no single method to investigate mediastinal LN invasion. Hence, a patient may have to undergo several tests and procedures. Noninvasive and invasive approaches are employed. Within the invasive techniques, endoscopic ultrasonography with needle aspiration (EUS-FNA) and endobronchial ultrasonography with transbronchial needle aspiration (EBUS-TBNA) are gaining importance in mediastinal staging.5 They provide ultrasonographic images and permit needle aspiration under direct vision for cytology specimen analysis. As more evidence is being accumulated on these staging approaches, the number of cervical mediastinoscopies, considered as the gold-standard for mediastinal staging, is diminishing.6

Characteristics of benign and malignant LNs using ultrasonography have been described in various contexts. Cervical and axillary LNs provided accurate characteristics (eg. shape, short- to long-axis ratio, number of blood vessels in LN, vascularization pattern, etc.) in predicting malignancy with linear superficial transducers.7-11 LN characteristics using EUS or EBUS also have established criteria predicting mediastinal LN malignancy (eg. size, shape, borders and echogenicity).12 Depending on the studies, it has been suggested to obtain specimens of all accessible LNs without considering their characteristics. It has also been suggested to proceed to a selective LN aspiration based on LN characteristics, with the advantage of cost reduction (fewer needles used, less time to carry out procedure, and specimens needed to be analysed).6

Color Doppler LN characteristics with endoluminal ultrasound (US) is only mentioned in a small number of studies and needs to be further investigated.13,14 With the good results obtained with superficial US, it seems reasonable to believe that color Doppler characteristics would increase accuracy in detecting malignancy of mediastinal LNs with endoluminal US.

New processors and probes are more accurate than the ones used in some of the past studies. Hence, the investigators can possibly obtain more precise findings than the ones the investigators can find in the literature.14

This study will consist of a prospective assessment of LN characteristics in patients undergoing EUS-FNA and/or EBUS-TBNA for diagnostic purposes. Cytology results will be considered as the gold-standard. By comparing the LN characteristics with the cytology results, the investigators will establish a scoring system to accurately predict malignancy.

The impact of this study is significant. If clinicians can accurately predict malignancy in mediastinal lymph nodes using ultrasound characteristics, biopsy of these lymph nodes could be avoided which would decrease the risk to the patient and the cost to the system (disposable needle costs, cytological preparation and analysis).

Hypotheses:

With a combination of endoluminal ultrasound characteristics, a simple scoring system can be established to help predict malignancy in mediastinal lymph nodes.

Objectives:

1. Establish a scoring system to accurately predict mediastinal lymph node malignancy with endoluminal ultrasound.
2. Retrospectively evaluate the impact of the established scoring system on the number of lymph nodes aspirations required for accurate staging.

Study Design:

Prospective, cohort study design. Clinical trial: Intervention - endoluminal ultrasound.

Methods:

This study will consist of a prospective non-randomized evaluation of endoluminal ultrasound characteristics in mediastinal lymph nodes using endoluminal ultrasound to predict malignancy within these nodes. All patients undergoing EUS-FNA and/or EBUS-TBNA for mediastinal LN staging for any suspected or confirmed malignancy at the CHUM - Hôpital Notre-Dame will be approached in an attempt to enroll them in the study. Patients will be enrolled and consented for the study during the pre-operative evaluation in the pre-operative clinic. The investigators will aim to recruit 100 consecutive patients.

Consented patients will undergo EUS with or without FNA and/or EBUS with or without TBNA in the same way as planned or decided during the procedure by the surgeon. During the procedure, data will be collected, including lymph node size, shape, border, echogenicity, homogeneity, location, color Doppler characteristics, number of nodes, etc. This will not add additional steps or time to the procedure. All this data and the cytology results obtained from EUS-FNA and EBUS-TBNA will be entered in a prospective database.

The cytology results will be considered as the gold-standard and with the collected characteristics univariate and multivariate logistic regressions will be used to establish a scoring system to predict malignancy. Sensitivity, specificity, positive predictive value, negative predictive value and accuracy will be determined based on the developed model.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing EUS-FNA and/or EBUS-TBNA for mediastinal LN assessment

Exclusion Criteria:

* Age < 18 years old
* Inability to consent to the study
* Medications including Warfarin (Coumadin) or Clopidogrel (Plavix)
* Coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 184 (Actual)
Dates: Start 2011-01; Primary Completion 2016-12 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
With a combination of endoluminal ultrasound characteristics, a simple scoring system can be established to help predict malignancy in mediastinal lymph nodes. | 3 months
  collected characteristics univariate and multivariate logistic regressions will be used to establish a scoring system to predict malignancy. Sensitivity, specificity, positive predictive value, negative predictive value and accuracy will be determined based on the developed model.

CONTACTS AND LOCATIONS:
Overall Officials: Moishe Liberman, MD, PhD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada